CLINICAL TRIAL: NCT01882725
Title: An Evaluation of the Effect of the Erchonia HP Scanner (HPS) Laser on Increasing Blood Circulation in Individuals With Chronic Heel Pain
Brief Title: Study of Low Level Laser Light Therapy to Improve Blood Circulation in People With Chronic Heel Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC_HPBC_001_ZANG
Record Dates: First submitted 2013-06-17; First posted 2013-06-20 (Estimated); Results first posted 2015-07-14 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Defective; Circulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erchonia HP Scanner (HPS) (Experimental): The Erchonia HP Scanner (HPS) Laser contains 3 independent diodes mounted in scanner devices and positioned equidistant from each other and titled at a 30 degree angle. Each scanner emits 17 milliwatts (mW), 635 nm of red laser light.
  Interventions: Device: Erchonia HP Scanner (HPS)

INTERVENTIONS:
Device: Erchonia HP Scanner (HPS) — The Erchonia HP Scanner (HPS) Laser is administered to the subject's heel 6 times across 3 consecutive weeks, 2 times each week, for 10 minutes of treatment time per administration.

SUMMARY:
The purpose of this study is to determine whether low level laser light therapy is effective in increasing local blood circulation in people with chronic heel pain arising from plantar fasciitis.

DETAILED DESCRIPTION:
Healthy blood circulation is important to overall health and well-being, as strong and steady local blood flow delivers fresh nutrients to the cells and prevents accumulation of waste materials within the cells necessary to maintain healthy cell function. Conversely, poor local blood circulation can cause numerous acute and chronic health problems, and can manifest itself in symptoms of pain, numbness, weakness and swelling, and can exacerbate these symptoms in co-existing acute and chronic conditions. Chronic conditions that may result from poor blood circulation that is untreated and persists over a long period of time include varicose veins, kidney damage, stroke and heart attack. Memory loss, frequent headaches, dizzy spells and slowed mental response can also result.

Therefore, improving local blood circulation has significant positive implications for both the overall health and well-being of an individual and for improving, relieving and preventing symptoms and long-term complications of poor blood circulation. Treatment to improve blood circulation include simple options such as changes in dietary and exercise habits, and alternative treatments such as acupuncture and herbal remedies. Medications may be prescribed to assist with contributory conditions such as high blood pressure or cholesterol. In more progressed cases, surgical options such as angioplasty or bypass may be performed to treat narrowed or blocked arteries.

However, less invasive options are usually minimally effective, medication has its own risks and side-effects and surgical procedures are invasive and carry significant procedural risks and potential complications. The purpose of this study is to evaluate the efficacy of low level laser therapy as a means of increasing local blood circulation as it is related to reducing chronic heel pain arising from plantar fasciitis that is simple, non-invasive and risk-free.

Low level laser therapy is believed to effect various physiological mechanisms of change that include improved blood flow and increased cell metabolism, advanced healing, anti-inflammatory actions and stimulation of the immune system. The laser directs light energy into the body's cells. The cells then convert this light energy into chemical energy to promote natural healing and pain relief. The laser also allows photons to enter the tissue and become absorbed in the cells mitochondria within which the photonic energy is converted to electromagnetic energy in the form of adenosine triphosphate (ATP). This additional ATP is energy the cell uses to trigger positive physiological responses from the body such as increased cell metabolism and development of muscle tissue and collagen, improvement of blood circulation, stimulation of tissue repair, wound healing and stimulation of the nervous and immune systems.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral Mechanical Plantar Heel Pain: insertional heel pain of the plantar fascia - plantar fasciitis - in one heel
* Chronic heel pain defined as at least 3 months of ongoing heel pain with no evidence of acute trauma to the heel
* A self-rating on the 0-100 Visual Analog Scale of at least 50 for heel pain experienced upon taking the first few steps of the study qualification evaluation day (recorded retrospectively), to be confirmed by the two-day average VAS attained during the Baseline Washout phase.
* Heel pain has been previously unresponsive to prescription non-steroidal anti-inflammatory drugs (NSAIDs) taken over a minimum period of 2 weeks; and any two or more of the following conservative treatments: rest, taping, stretching, orthotics, shoe modifications, night splinting, casting, physical therapy, or local corticosteroid injections.
* Subject is willing and able to refrain from consuming over-the-counter and/or prescription medications for the indication of the relief of pain throughout the study.
* Subject is willing and able to refrain from partaking in other non-study treatments or therapies for the relief of heel pain throughout the study.

Exclusion Criteria:

* Subject does not have any one or more of the following etiologies of chronic heel pain: Mechanical Posterior Heel Pain; Neurologic Heel Pain; Arthritic Heel Pain; and Traumatic Heel Pain
* Evidence of acute trauma to the heel
* Loss of plantar foot sensation
* Foot deformity
* Previous surgery to the heel
* Foot trauma within the previous three months
* Skin ulceration - infection or wound - on the heel and surrounding treatment area
* Sciatica
* Benign and malignant tumors
* Acute infection of soft tissue/bone, e.g. osteomyelitis
* Presence of diabetic neuropathic pain
* Diabetes Type I
* Presence of sensory neuropathy
* Previous diagnosis of neuropathy affecting lower extremities
* Peripheral vascular disease or autoimmune disease
* Fibromyalgia
* Chronic fatigue syndrome
* Chronic pain disorders
* Metabolic disorders: Osteomalacia, Paget's disease, Sickle cell disease
* Blood coagulation disorders
* Significant heart conditions including Congestive Heart Failure (CHF) and implantable heart devices
* Non-ambulatory status
* Unable or unwilling to consume the study rescue medication of Tylenol
* Photosensitivity disorder
* Pregnant or lactating
* Serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in past two years
* Developmental disability or cognitive impairment that would preclude adequate comprehension of the consent form and ability to record the necessary measurements.
* History of drug or alcohol abuse
* Involvement in litigation and/or a worker's compensation claim and/or receiving disability benefits related to the study condition
* Participation in any type of research in the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Zang, DPM, Principal Investigator
Locations (1):
- Arizona Institute of Footcare Physicians, Mesa, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erchonia HP Scanner (HPS)
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Erchonia HP Scanner (HPS)
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.79 (11.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14
Duration of Heel Pain [Mean (Standard Deviation); unit: months] — Duration of heel pain is recorded as number of months of chronic heel pain experienced prior to study enrollment
  months | 15.93 (15.52)
Degree of Heel Pain on the Visual Analog Scale (VAS) [Mean (Standard Deviation); unit: units on a scale] — The Visual Analog Pain Scale (VAS) is one of the three most commonly used scales for assessing chronic pain consisting of a 100 millimeter (mm) horizontal line anchored at one end by the label "0: no pain at all" and at the other end "100: worst pain imaginable". The subject marks on the line the spot for the overall degree of pain experienced in the study treated heel region upon waking in the morning and taking the first few steps of the day, which is then measured using a ruler.
  units on a scale | 69.29 (10.67)

OUTCOME MEASURES:

1. Primary Outcome: Change in Skin Perfusion Pressure (SPP)
Description: Skin Perfusion Pressure (SPP) measured peripheral microcirculation or skin perfusion using a laser Doppler sensor and a pressure cuff to evaluate reactive hyperemia, the transient increase in blood flow that occurs following a brief period of ischemia. The SPP value was measured in mmHg.
  The per cent (%) change in mean Skin Perfusion Pressure (SPP) in mmHg was calculated as the % change in measurements from before the first procedure administration with the Erchonia® HPS Laser to after the sixth and final procedure administration. It was pre-determined that a minimum mean change in % SPP of +10% or greater across the evaluation period would be considered clinically meaningful.
  A positive (+) change indicates that SPP increased across the procedure administration phase and is positive for study efficacy.
  A negative (-) change indicates that SPP decreased across the procedure administration phase and is negative for study efficacy.
Time Frame: baseline and 3 weeks
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Erchonia HP Scanner (HPS)
Number analyzed (Participants) | 14
percentage of change | 17.68 (30.37)
Statistical Analysis 1: Comparison: Erchonia HP Scanner (HPS); Test type: Superiority or Other; p < 0.05, t-test, 1 sided

2. Secondary Outcome: Change in Skin Surface Temperature on the Hind Foot
Description: Skin surface temperature on the hind foot was recorded in degrees using an infrared thermometer. Change in skin surface temperature in degrees was calculated as the change in measurements before the first procedure administration (baseline) to after the sixth and final procedure administration. It was pre-determined that a minimum mean increase in skin surface temperature of +2.5 degrees across the procedure administration phase would be considered clinically meaningful.
  A positive (+) change indicates that the skin surface temperature increased across the procedure administration phase and is positive for study efficacy.
  A negative (-) change indicates that the skin surface temperature decreased across the procedure administration phase and is negative for study efficacy.
Time Frame: baseline and 3 weeks
Measure: Mean (Standard Deviation); unit: Degrees Farenheit
Arm/Group | Erchonia HP Scanner (HPS)
Number analyzed (Participants) | 14
Degrees Farenheit | 2.93 (3.55)
Statistical Analysis 1: Comparison: Erchonia HP Scanner (HPS); Test type: Superiority or Other; p < 0.01, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Erchonia HP Scanner (HPS)
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No